CLINICAL TRIAL: NCT06306820
Title: Ultrasound Guided Recruitment Manauvere Versus Individualized Positive End Expiratory Pressure in Pediatric Patients Undergoing Laparoscopic Abdominal Surgery; A Prospective Randomized Controlled Study.
Brief Title: Ultrasound Guided Recruitment Manauvere Versus Individualized Positive End Expiratory Pressure in Pediatric Patients Undergoing Laparoscopic Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reham Mostafa Mostafa Rezk, Principal Investigator of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264MS257/7/2023
Record Dates: First submitted 2024-03-02; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Ultrasound Guided Recruitment Manauvere; End Expiratory Pressure; Pediatric Patients; Laparoscopic Abdominal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients will receive a fixed positive end-expiratory pressure (PEEP) of 5 cmH2O.
  Interventions: Other: Fixed PEEP
- Ultrasound group (Experimental): Patients will receive ultrasound -guided lung recruitment.
  Interventions: Other: Ultrasound-guided lung recruitment
- PEEP IND group (Experimental): Patients will receive individualized positive end-expiratory pressure (PEEP).
  Interventions: Other: Individualized PEEP

INTERVENTIONS:
Other: Fixed PEEP — Patients will receive a fixed positive end-expiratory pressure (PEEP) of 5 cmH2O throughout the surgical procedure.
  Arms: Control group
Other: Ultrasound-guided lung recruitment — Patients will receive ultrasound-guided lung before pneumoperitoneum, after pneumoperitoneum then once an hour, until the end of surgery. Alveolar recruitment will be conducted the same as that for the conventional manoeuvre with a simultaneous continuous ultrasound assessment if atalectasis is detected until no collapsed areas are visualized. When the collapsed lung areas are absent on the sonogram, positive end-expiratory pressure (PEEP) can no longer increase at this point. Subsequently, the pressure will be maintained for approximately 10 breaths.
  Arms: Ultrasound group
Other: Individualized PEEP — Patients will receive individualized positive end-expiratory pressure (PEEP). After the first recruitment Maneuvere (RM), titration of PEEP will be performed by setting the initial PEEP to 5 cm H2O, then increasing PEEP according to the gradient of 2 cmH2O every 3 min, calculating static compliance (Cstat) according to the formula: [Cstat = VT/Pplat - PEEP] (Pplat = plateau pressure), then gradually increasing PEEP, until the calculated Cstat shows a downward trend, the we set its previous PEEP (corresponding to PEEP for high Cstat) as the optimal PEEP for this patient. The highest PEEP is limited to 15 cmH2O.
  Arms: PEEP IND group

SUMMARY:
The aim of this prospective randomized controlled study is to compare the effect of US-guided Recruitment Manauvere (RM) versus individualized positive end-expiratory pressure (PEEP) on oxygenation and preventing respiratory complications in pediatric patients undergoing laparoscopic abdominal surgeries.

DETAILED DESCRIPTION:
Atelectasis is among the most frequent postoperative pulmonary complications (PPCs) of general anesthesia with an incidence of between 68% and 100% in children. Atelectasis impairs gas exchange, thus causing hypoxemia and other respiratory disorders such as acute lung injury and pneumonia.

Pneumoperitoneum is another risk factor for perioperative atelectasis. It elevates the diaphragm and intra-abdominal pressure. In order to prevent atelectasis, applying positive end-expiratory pressure (PEEP) or an alveolar recruitment Maneuvere (RM) have shown beneficial effects.

Lung ultrasound (US) is a noninvasive, radiation-free, convenient, and reproducible bedside imaging modality for anesthesia-induced atelectasis in children.

ELIGIBILITY:
Inclusion Criteria:

* Age from 3 to 8 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Children scheduled for elective laparoscopic abdominal surgeries.

Exclusion Criteria:

* Parental refusal.
* Bronchial asthma or any preexisting chest disease.
* Congenital deformity of the thoracic cage.
* Patients with a history of thoracic surgery.
* Cardiac, hepatic, or renal failure.
* Obese children with BMI at or above 95th percentile of the same age and sex.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative oxygenation | One hour after second recruitment Maneuvere
  Intraoperative oxygenation which will be assessed by P/F ratio (the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen P/F ratio will be assessed before induction of anesthesia, one hour after pneumoperitoneum, and after second recruitment Maneuvere (RM)

SECONDARY OUTCOMES:
Lung ultrasound scores | 24 hours after extubation
  Lung ultrasound scores to assess anesthesia-induced atelectasis and will be performed immediately after intubation, one hour after pneumoperitoneum, one hour after extubation, and 24 hours after extubation
Mean arterial blood pressure (MAP) | One hour after extubation
  Mean arterial blood pressure (MAP) will be assessed before induction of anesthesia, immediately after intubation, after first recruitment Maneuvere (RM), one hour after pneumoperitoneum, after second recruitment Maneuvere (RM), and one hour after extubation.
Heart rate | One hour after extubation
  Heart rate (HR) will be assessed before induction of anesthesia, immediately after intubation, after first recruitment Maneuvere (RM), one hour after pneumoperitoneum, after second recruitment Maneuvere (RM), and one hour after extubation.
Postoperative pulmonary complication | 24 hours postoperative
  Early postoperative pulmonary complication in the first 24 hours postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.